CLINICAL TRIAL: NCT07374601
Title: The Predictive Value of Super-resolution Ultrasound Microvascular Imaging for the Prognosis of Peripheral Artery Disease
Brief Title: The Value of Super-resolution Ultrasound Imaging for Peripheral Artery Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Xinzhi Yang, Clinical Professor, Peking University First Hospital
Other Study IDs: 2025R0004
Record Dates: First submitted 2026-01-12; First posted 2026-01-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 300 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy People
- PAD Patients

SUMMARY:
Peripheral artery disease (PAD) is a chronic atherosclerotic disorder characterized by stenosis or occlusion of the extracranial arteries distal to the aortic arch, most commonly affecting the lower extremities. This vascular compromise leads to tissue hypoperfusion, resulting in a spectrum of clinical manifestations ranging from asymptomatic disease to intermittent claudication, critical limb ischemia, and limb loss.

The microvascular system comprises arterioles, capillaries, and post-capillary venules with diameters less than or equal to 100 micrometers. Emerging evidence underscores that microvascular dysfunction (MVD)-defined as structural and functional impairment of this microcirculatory network-plays a pivotal pathophysiological role in PAD progression, contributing to impaired perfusion reserve, endothelial dysfunction, inflammation, and tissue fibrosis, independent of macrovascular stenosis severity.

Super-resolution ultrasound microvascular imaging (SRUMI) is an advanced contrast-enhanced ultrasound technique that leverages the nonlinear acoustic signatures of intravascular microbubble contrast agents (e.g., SonoVue) under ultra-low mechanical index (MI) pulsing schemes. Implemented on the Verasonics Vantage 256 research platform (Verasonics, Inc., Kirkland, WA, USA), SRUMI achieves in vivo visualization of microvascular architecture at sub-diffraction resolution (approximately 10-20 micrometers), surpassing conventional Doppler and contrast-enhanced ultrasound. Key advantages include absence of ionizing radiation, negligible thermal and mechanical bioeffects, real-time capability, portability, and cost-effectiveness. As such, SRUMI represents a promising noninvasive tool to probe microvascular integrity in PAD, enabling mechanistic investigation of MVD's contribution to disease initiation, progression, and therapeutic response.

This study aims to evaluate the diagnostic and prognostic utility of SRUMI for assessing microvascular dysfunction in patients with PAD. The investigators prospectively enrolled patients diagnosed with PAD and admitted to the Department of Interventional Vascular Surgery at Peking University First Hospital. Primary objectives include:

Characterizing lower-limb microvascular density, morphology, and perfusion patterns via SRUMI across PAD subgroups stratified by comorbidities-including diabetes mellitus, current or former smoking, hypertension, and chronic kidney disease;

Assessing the concordance between SRUMI-derived microvascular parameters and established clinical and paraclinical markers, including symptom severity (Rutherford classification), ankle-brachial index (ABI), urinary albumin-to-creatinine ratio (UACR), and retinal microvascular findings on fundoscopy;

Determining the sensitivity, specificity, and predictive value of baseline SRUMI metrics for major adverse limb events (MALE) and cardiovascular outcomes during longitudinal follow-up; and

Comparing the incremental prognostic value of SRUMI against conventional modalities-including ABI, duplex ultrasonography, and clinical risk scores-using multivariable Cox regression and time-dependent receiver operating characteristic (ROC) analyses.

Collectively, this research seeks to establish SRUMI as a quantitative, translatable biomarker of microvascular health in PAD, thereby advancing precision phenotyping, risk stratification, and monitoring of therapeutic efficacy in this high-morbidity population.

ELIGIBILITY:
*Inclusion Criteria:*

1. Adults aged ≥18 years and ≤100 years;
2. Diagnosis of peripheral artery disease (PAD) confirmed by comprehensive clinical assessment-including characteristic symptoms (e.g., intermittent claudication, rest pain), physical findings (e.g., diminished or absent distal pulses, bruits), ankle-brachial index (ABI) < 0.9, and corroborating vascular imaging (e.g., duplex ultrasonography, CTA, or MRA);
3. Alternatively, healthy adults without PAD (i.e., ABI ≥ 0.9, absence of suggestive symptoms or signs, and no history of atherosclerotic cardiovascular disease) who meet all other eligibility requirements;
4. Willing and able to provide written informed consent.

*Exclusion Criteria:*

1. Inability to complete study procedures due to:

   1. Severe involuntary movement disorders (e.g., advanced Parkinson's disease or cerebellar ataxia) interfering with image acquisition;
   2. Contraindication to contrast-enhanced ultrasound (e.g., documented hypersensitivity to sulfur hexafluoride microbubble contrast agent [SonoVue®]);
   3. Active lower-limb infection (e.g., diabetic foot infection with systemic signs or osteomyelitis), which precludes safe or interpretable data collection;
2. Cognitive impairment or legal incapacity precluding autonomous informed consent;
3. Refusal-by the participant or their legally authorized representative-to provide informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: **Study Population Description:** Participants will be recruited from the Department of Interventional Vascular Surgery at Peking University First Hospital. The cohort comprises two parallel groups: (i) patients hospitalized with a confirmed diagnosis of PAD, and (ii) control participants without PAD (i.e., non-atherosclerotic controls), matched for age and sex where feasible. Enrollment adheres strictly to the prespecified inclusion and exclusion criteria above.
  **Sampling Method:** Convenience sampling (a form of non-probability sampling), reflecting real-world clinical recruitment within a single tertiary academic medical center.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01-08 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
microvascular density | Baseline; Perioperative(before endovascular surgery)

IPD SHARING:
Plan to Share IPD: No